CLINICAL TRIAL: NCT00102505
Title: Phase I Trial of Motexafin Gadolinium (MGd) in Combination With Docetaxel and Cisplatin for Treatment of Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Motexafin Gadolinium (MGd) in Combination With Docetaxel and Cisplatin for Treatment of Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0220
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Non-Small-Cell Lung Carcinoma; Carcinoma, Bronchogenic
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; Metastatic lung cancer; Inoperable lung cancer; Advanced lung cancer; Large-cell lung cancer; Adenocarcinoma, lung; Squamous cell carcinoma, lung; Squamous cell lung cancer; Large cell carcinoma, lung; Bronchogenic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Bronchogenic; Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Squamous Cell; Carcinoma, Large Cell | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: Motexafin Gadolinium Injection

SUMMARY:
The purpose of the study is to determine the dose limiting toxicities and maximum tolerated dose of motexafin gadolinium when administered with docetaxel and cisplatin in patients with Non-small Cell Lung Cancer.

A cycle consists of 3 weeks. During week 1, patients receive MGd, docetaxel, and cisplatin treatment followed by 2 weeks without treatment.

Eligible patients will receive 1 or 2 doses of MGd, depending on cohort, and a single dose of docetaxel and cisplatin at 75 mg/m² during the first week of each cycle. Additionally, tumor response will be evaluated at the end of even numbered cycles (2, 4, and 6). Patients may stay on the study a maximum of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* ECOG score of 0, 1, or 2
* Histologically confirmed diagnosis of non-small cell lung cancer

Exclusion Criteria:

Laboratory values demonstrating inadequate function of the following:

* Bone marrow
* Kidneys
* Liver

and

* Peripheral neuropathy Grade 2 or higher
* Greater than 2 prior chemotherapy regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2004-11

PRIMARY OUTCOMES:
Dose limiting toxicities of MGd when administered concurrently with docetaxel and cisplatin
Maximum tolerated dose of MGd when administered concurrently with docetaxel and cisplatin

SECONDARY OUTCOMES:
Tumor response

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States